CLINICAL TRIAL: NCT04707924
Title: Within-subject, Investigator Initiated, Single-blind, Single-centre, Randomized Clinical Trial Investigating the Efficacy of Fractional Er:YAG Laser in Lupus Erythematosus Scars
Brief Title: Efficacy of Fractional Er:YAG Laser in Lupus Erythematosus Scars
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to enroll patients
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-00987
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Lupus Erythematosus, Cutaneous
Keywords: Lupus; Laser; CO2; Er:YAG
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: 1:1 within-subject random allocation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Er:YAG laser (Experimental): Treatment of scars with fractional Er:YAG 2940nm laser.
  Interventions: Device: Er:YAG laser
- Control area (No Intervention): No treatment performed on control areas.

INTERVENTIONS:
Device: Er:YAG laser — Treatment of scars with fractional Er:YAG 2940nm laser.
  Arms: Er:YAG laser

SUMMARY:
Cutaneous Lupus erythematosus (CLE) is a chronic autoimmune connective tissue disease with a prevalence of 14.6 - 73.2/100,000, predominantly in women in mid adulthood. Cutaneous lesions occur in about 75-80% of patients with systemic lupus erythematodes.These lesions unfortunately and invariably lead to significant scarring and postinflammatory hypo- and hyperpigmentation.

Several studies have reported that laser treatments in patients with CLE have a positive effect and safety. However, only few case reports exist about the effect of ablative lasers such as Carbon Dioxide (CO2) and Erbium-doped Yttrium Aluminum Garnet (Er:YAG) lasers in CLE scarring.

Although no study shows a flare-up of CLE after laser treatment of the scars, many physicians are afraid of treating these often stigmatizing scars. Considering the huge psychological impact of facial scaring on quality of life, it is essential to explore and assess the value of already well-established treatment options for the management of scars also in patients with cutaneous lupus erythematodes.

Hereby the study seeks the subjective and objective improvement of the CLE-scars after treatment with fractional Er:YAG laser compared to control (untreated) areas.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Skin type I-IV
* Presence of >1 scar due to CLE at one localisation
* Stable disease (without or with permanent therapy >3months)

Exclusion Criteria:

* History of adverse events related to ablative fractional laser therapy
* Ablative resurfacing within the last 6 months on the scar
* Pregnant or breast feeding women
* Intake of isotretinoin in the last 6 month
* Intention to become pregnant during the course of the study
* Any scar treatment in the last 3 month before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Average reduction of POSAS scar severity measure. | 24 weeks
  Average reduction from baseline of Patient and Observer Scar Assessment Scale (POSAS), ranging from 12 to 120 with higher score indicating a worst condition.

SECONDARY OUTCOMES:
Cumulative incidence of localized disease flare-up. | 4, 8, 12, 16 and 24 weeks
  Cumulative incidence of disease flare-up defined according to localized Revised Cutaneous Lupus Erythematosus Disease Area and Severity Index (RCLASI) difference from baseline of 1 point or above. The localized RCLASI ranges from 0 to 13, with higher scores indicating a worst local disease activity.
Overall average reduction of POSAS scar severity measure. | 16 and 24 weeks
  Overall average reduction from baseline of Patient and Observer Scar Assessment Scale (POSAS), ranging from 12 to 120 with higher score indicating a worst condition.
Overall average scar improvement according to physician global assessment. | 4, 8, 12, 16 and 24 weeks
  Overall average scar improvement from baseline according to a 6-point Physician Global Assessment (PGA) scale, based on before-after pictures of lesions assessment, ranging from 1 to 6, with higher scores indicating a better outcome.
Average patient's satisfaction. | 16 and 24 weeks
  Average patient's satisfaction score as assessed by a 9-point anchored visual analogue scale (VAS), ranging from -4 to +4, with negative scores indicating a worsening of condition compared to the untreated control scar, with 0 indicating no difference and with positive scores indicating an improvement.

OTHER OUTCOMES:
Proportion of observed side-effects. | 24 weeks
  Proportion of observed treatment side-effects, such as hyperpigmentation and erythema.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Heidemeyer, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Department of dermatology, University Hospital Inselspital, Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No